CLINICAL TRIAL: NCT05218538
Title: Liver Cirrhosis Diagnosis Prioritizing Algorithm Based on Electronic Health Records.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Ziv Neeman, Director of Imaging Institute & Nuclear Medicine, HaEmek Medical Center, Israel
Other Study IDs: 0208-20-EMC
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: NAFLD - Nonalcoholic Fatty Liver Disease; Fibrosis, Liver; Cirrhosis, Liver
Keywords: Fibroscan; Model; Machine learning
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Learning e-cohort: Includes the entire population within Clalit Healthcare's electronic records database which spans from the year 2000 to 2021.
- FIB-4 score group: One of the two validation population invited to the clinic. The FIB-4 score group are individuals invited by their score.
  Interventions: Diagnostic Test: Fibroscan (non interventional)
- Model based group: One of the two validation population invited to the clinic:
  The Model based group are individuals invited by their predicted time-to-event to liver cirrhosis diagnosis.
  Interventions: Diagnostic Test: Fibroscan (non interventional)

INTERVENTIONS:
Diagnostic Test: Fibroscan (non interventional) — An elastography test that includes an ultrasound wave imaging of the liver to estimate liver fatness, in combination with a proprioty examination of the liver stiffness.
  Groups: FIB-4 score group; Model based group

SUMMARY:
The investigators use machine learning capabilities on massive electronic health records for the purpose of developing a model that prioritizes individuals at high risk of progressing to liver cirrhosis, and validating it with participants that the model found to be at high risk.

constructing and validating a reliable model, with sufficient accuracy to justify further and expensive means of detection, will enable treating patients with damaged liver at an early enough stage to allow improvement of the liver condition.

DETAILED DESCRIPTION:
In this study the investigators harness modern capabilities of machine learning in the field of hepatology for developing a model that can identify prioritize individuals at high risk of progressing to liver cirrhosis at an early and treatable stage.

Cirrhosis is an advanced state of liver disease that usually manifest when the liver is already severely damaged, without many treatment options and gloomy prognosis.

There are currently 2 means for diagnosis, the first is liver biopsy that is costly and inflicts pain to the patients, and has its own risks. The second is a designated imaging test, such as Fibroscan, which is safe and painless but also too expensive than can be doable as a broad screening tool.

Scores that calculates higher probability for a liver disease have already been developed, but with lower predictive strength than suitable to justify further examination towards detection.

The study comprises of 4 distinct phases:

1. Model development. A machine learning model predicting time-to-event for liver cirrhosis diagnosis will be developed based on Electronic Health Records. Records are anonymized and all work is performed on a designated server.
2. Anonymized Electronic Health Records latest lab test results and diagnoses from Clalit healthcare's North district will be obtained. On those records the trained model from phase 1 will run to predict time-to-event for liver cirrhosis diagnosis. Via predictions individuals will be ordered by risk.

   Via the deanonymized records, available only to clinicians, 20 individuals of highest risk will be observed. This includes measuring latest FIB-4 scores, viewing prior diagnoses and tests, as well as textual information from physicians. These individuals are not invited to a visit and are only viewed retrospectively through their records.
3. Upon results from phase 2 the machine learning model from phase 1 will be revised. This includes possible alterations such as revisions of inclusion/exclusion criteria, change of lab tests given as input to the model, etc.
4. As in phase 2, updated anonymized Electronic Health Records from Clalit healthcare's North district will be obtained. The updated model from phase 3 will run to predict time-to-event for liver cirrhosis diagnosis. In addition, all individuals will have their FIB-4 score computed. A ranked list of the top individuals with highest predicted risk predicted by the model from phase 3 and top individuals with the highest FIB-4 score will be constructed. Approximately a fourth of the individuals will come from the FIB-4 score group, age and gender matched to the prediction group. Group identity will remain unknown to clinicians, maintaining a double blinded study. Individuals will be invited to the clinic for checks. At the clinic individuals will undergo Fibroscan, height and weight measurements, answer the WHO Alcohol Use Disorders Identification Test (AUDIT) questionnaire. Furthermore, their files within the Electronic Health Records will be open and existing diagnoses, lab tests and medication prescriptions be collected.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with electronic health records from Clalit Healthcare's North district
* Ages 40-75

Exclusion Criteria:

* No lab test results for Hemoglobin, platelet, or white blood cell count.
* Known Viral Hepatitis (HBV, HCV, HDV).
* Known liver cirrhosis.
* Known lipidoses.
* Known alpha-1-antitrypsin deficiency.
* Known hemochromatosis.
* Known disorders of copper metabolism.
* Known Budd-Chiari syndrome.
* Known alcoholic fatty liver.
* Known diagnosis for alcohol abuse.
* Known Autoimmune Hepatitis.
* Known biliary cirrhosis.
* Known cholangitis.
* Undergone liver replacement by transplant.
* Right Heart Failure.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study has two main populations:
  * The entire population within Clalit Healthcare's electronic records database.
  * Community based healthy subjects without known viral or autoimmune hepatitis, and without right heart failure.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of advanced liver fibrosis by Fibroscan (kPa measure as a grade between F3-F4). | 6 - 12 months
  measurement ranges from a min value of 0 to a max value of 75. For NAFLD above 7.5 is considered F2,above 10 F3 and above 14 high.

SECONDARY OUTCOMES:
Abnormal liver Fibroscan (kPa measure as a grade between F1-F2). | 6 - 12 months
  measurement ranges from a min value of 0 to a max value of 75. For NAFLD above 7.5 is considered F2,above 10 F3 and above 14 high.
Fatty liver (score as measured in CAP) | 6 - 12 months
  measurement ranges from a min value of 100 to a max value of 400. Above 290 is considered high.

CONTACTS AND LOCATIONS:
Overall Officials: Ziv Neeman, MD, Principal Investigator — HaEmek Medical Center, Israel
Locations (1):
- Haemek medical center, Afula, North, Israel

REFERENCES:
- [Derived] Kalka IN, Hazzan R, Yacovzada NS, Igbaria S, Segal E, Weinberger A, Neeman Z. Fibro predict a machine learning risk score for advanced liver fibrosis in the general population using Israeli electronic health records. Sci Rep. 2025 Sep 1;15(1):32035. doi: 10.1038/s41598-025-17534-9. PMID 40887472